CLINICAL TRIAL: NCT05898594
Title: Evaluating the Feasibility of Lung Cancer Screening in High-risk Black Individuals
Brief Title: Lung Cancer Screening in High-risk Black Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chi-Fu Jeffrey Yang, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-382; 1R18HS029430-01 (AHRQ)
Record Dates: First submitted 2023-05-26; First posted 2023-06-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; Lung Carcinoma
Keywords: Lung Cancer; Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening: Low-Dose Computed Tomography Screening (Experimental): Participants will undergo study procedures as outlined:
  * Complete questionnaires pre- and post- low-dose computed tomography (LDCT) test.
  * Visit Massachusetts General Hospital facility for a LDCT screening test.
  Interventions: Procedure: Low-dose Computed Tomography

INTERVENTIONS:
Procedure: Low-dose Computed Tomography — Per standard care

SUMMARY:
The goal of this research study is to study U.S. Black individuals with a history of smoking to examine the feasibility, acceptability, and performance of low-dose computed tomography (LDCT) screening among this population.

The name of the intervention used in this research study is:

Low-dose computed tomography (radiologic scan) chest scan

DETAILED DESCRIPTION:
The goal of this single-arm pilot research study is to evaluate the feasibility and acceptability of low-dose computed tomography (LDCT) screening for lung cancer among U.S. Black individuals with a history of smoking.

LDCT screening is currently the only recommended way to screen for lung cancer among high-risk individuals. However, many Black individuals at high-risk for lunch cancer are currently ineligible for lung cancer screening.

Study procedures include screening for eligibility, completion of questionnaires, and a LDCT screening test.

Participation in this study is expected to last up to 3 months.

It is expected about 900 people will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Black individual.
* Have a self-reported history of smoking. No restriction will be placed on the number of smoking pack years participants must have nor the number of years former smokers must have quit smoking.
* Aged >= 50 years.

Exclusion Criteria:

* Individuals with a history of lung cancer.
* Individuals with symptoms suggestive of lung cancer. We will evaluate whether individuals have symptoms suggestive of lung cancer by administering an online screening questionnaire, which will ask whether they have experienced shortness of breath, whether they become easily winded, and whether they have had a chronic cough within the last 12 weeks that has not improved. Individuals who select that they have any one of these symptoms will be advised to follow up with their primary doctor and will not be eligible to participate in the study.
* Individuals with pneumonia or acute respiratory infection within 12 weeks prior to enrollment that was treated with antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 900 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Enrolled Participants | At enrollment
  Primary endpoint is feasibility. Feasibility is defined as the percentage of individuals invited to participate in the trial who enroll.
Proportion of Participants with Positive Low-dose Computed Tomography Test | At 3 months
  The percentage of participants who have a positive low-dose computed tomography test will be evaluated. This percentage will be compared to the Black individuals randomized to the low-dose computed tomography screening arm in the National Lung Screening Trial (historical control).
Proportion of Participants Diagnosed with Invasive Lung Cancer | At 6 months
  The proportion of participants with a lung cancer diagnosis post-low-dose computed tomography screening test will be compared to Black individuals randomized to the LDCT screening arm in the National Lung Screening Trial (historical control).
Distribution of Lung Imaging Reporting and Data System (Lung-RADS) Scores | At 3 months
  The distribution of Lung-RADS scores among participants will be evaluated and compared to the distribution of Lung-RADS scores among Black individuals randomized to the LDCT screening arm in the National Lung Screening Trial (historical control).

SECONDARY OUTCOMES:
Proportion of Participants Who Undergo Invasive Diagnostic Procedures | At 6 months
  The proportion of participants who undergo invasive diagnostic procedures will be evaluated and compared to the proportion of Black individuals randomized to the LDCT screening arm in the National Lung Screening Trial (historical control) who underwent invasive diagnostic procedures.
Proportion of Participants Who Have a Complication Resulting from an Invasive Diagnostic Procedure Performed for a Positive Low-dose Computed Tomography Scan | At 6 months
  The proportion of participants who have a complication resulting from an invasive diagnostic procedure performed for a positive low-dose computed tomography scan will be evaluated. This proportion will be compared to the proportion of Black individuals randomized to the low-dose computed tomography screening arm in the National Lung Screening Trial (historical control) who had a complication resulting from an invasive diagnostic procedure performed for a positive low-dose computed tomography scan.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fu Jeffrey Yang, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation